CLINICAL TRIAL: NCT04318327
Title: Phase I, Open Label, Study of B-cell Maturation Antigen (BCMA)-Directed CAR-T Cells in Adult Patients With Multiple Myeloma
Brief Title: BCMA-directed CAR-T Cell Therapy in Adult Patients With Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CADPT07A12101
Record Dates: First submitted 2020-03-20; First posted 2020-03-23 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; B-cell maturation antigen; BCMA; anti-BCMA; BCMA-directed; chimeric antigen receptor; CAR-T; PHE885
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PHE885 (Part A) (Experimental): Relapsed and/or refractory multiple myeloma (r/r MM) patients will receive PHE885.
  Interventions: Biological: PHE885
- PHE885 (Part B) (Experimental): Newly diagnosed multiple myeloma (NDMM) patients will receive PHE885.
  Interventions: Biological: PHE885

INTERVENTIONS:
Biological: PHE885 — Infusion

SUMMARY:
This was a first-in-human study to evaluate the feasibility, safety and preliminary antitumor efficacy of autologous T cells genetically engineered with a novel B-cell Maturation Antigen (BCMA)-specific chimeric antigen receptor (CAR) and manufactured with a new process. CAR-T cells were investigated as a single agent in multiple myeloma

DETAILED DESCRIPTION:
This was a phase I, open label study to characterize the safety and tolerability of a novel B-cell Maturation Antigen (BCMA)-specific chimeric antigen receptor (CAR) manufactured with a new process. In the dose escalation part (Part A) of the study, the anti-BCMA CAR-T cell therapy was studied in adult multiple myeloma (MM) subjects who were relapsed and/or refractory. In the dose evaluation part (Part B) of the study, the anti-BCMA CAR-T cell therapy was studied in newly diagnosed adult subject with MM.

ELIGIBILITY:
Inclusion Criteria:

* Part A: Subjects with MM who are relapsed and/or refractory to at least 2 prior treatment regimens, including an IMiD (e.g. lenalidomide or pomalidomide), a proteasome inhibitor (e.g. bortezomib, carfilzomib), and an approved anti-CD38 antibody (e.g. daratumumab), if available, and have documented evidence of disease progression (IMWG criteria)
* Part A: ECOG performance status that is either 0 or 1 at screening
* Part B: Subjects with newly diagnosed multiple myeloma (NDMM) who have received a minimum of 4 and up to 6 cycles of standard induction therapy with VRd, D-VRd, or D-Rd, and have achieved a response of PR or better. One cycle of CyBorDex is allowed prior to induction.
* Part B: ECOG performance status that is either 0,1 or 2 at screening
* Measurable disease as defined by the protocol
* Adequate hematological values
* Must have a leukapheresis material of non-mobilized cells accepted for manufacturing

Exclusion Criteria:

* Prior administration of a genetically modified cellular product including prior BCMA CAR-T therapy. Patients who have received prior BCMA-directed bi-specific antibodies or antibody-drug conjugates (ADC) are not excluded.
* Autologous HSCT within 6 weeks prior to enrollment or any prior history of allogeneic hematopoietic stem cell transplant (HSCT)
* Chemotherapy or any concomitant anti-cancer therapies (other than protocol prescribed lymphodepletion (LD) chemotherapy) within 2 weeks prior to apheresis
* Treatment with small molecule targeted antineoplastics within 2 weeks of apheresis collection or 5 half-lives whichever is shorter
* Have received antibodies or immunotherapies (other than daratumumab) within 4 weeks prior to apheresis collection. Daratumumab within 3 weeks prior to apheresis collection.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose limiting toxicities (DLT) | 28 days
  Incidence of Dose Limiting Toxicities (DLTs) during the first 28 days after anti-BCMA CAR-T cell administration
Nature of Dose limiting toxicities (DLT) | 28 days
  Nature of Dose Limiting Toxicities (DLTs) during the first 28 days after anti-BCMA CAR-T cell administration
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | 24 months

SECONDARY OUTCOMES:
Manufacture success rate (defined as number of subjects treated with planned target dose divided by total number of subjects treated) | 24 Months
  evaluate the feasibility of the manufacturing process
Overall Response Rate (ORR) in Part A | 24 months
  Proportion of subjects with the best overall response (BOR) of PR (partial response) or better, as determined by local investigator using the IMWG Criteria
ORR in Part B | 24 months
  Proportion of subjects with VGPR (very good partial response) or PR to induction therapy who achieve the BOR of PR or better, as determined by local investigator using the IMWG Criteria
Response rate at 3 and 6 months in Part A | 3 months, 6 months
  Proportion of subjects with the overall response of PR or better at months 3 and 6 after infusion respectively, as determined by local investigator using the IMWG Criteria
Overall response rate at 3 and 6 months in Part B | 3 months, 6 months
  Proportion of subjects with VGPR or PR to induction therapy who achieve the overall response of PR or better at months 3 and 6 after infusion respectively, as determined by local investigator using the IMWG Criteria
Overall Complete Response Rate (CRR) in Part A | 24 months
  Proportion of subjects with the BOR of CR or better, as determined by local investigator using the IMWG Criteria
Overall CRR in Part B | 24 months
  Proportion of subjects with a response of VGPR or PR to induction therapy with the BOR of CR or better, as determined by local investigator using the IMWG Criteria
CRR at months 3 and 6 in Part A | 3 months, 6 months
  Proportion of subjects with the overall response of CR or better at months 3 and 6 respectively, as determined by local investigator using the IMWG Criteria
CRR at months 3 and 6 in Part B | 3 months, 6 months
  Proportion of subjects with a response of VGPR or PR to induction therapy with the overall response of CR or better at months 3 and 6 after infusion, respectively, as determined by local investigator using the IMWG Criteria
DOR (duration of response) in Part A | from disease response to disease progression, assessed up to approximately 24 months
  DOR as assessed by local investigator: the time from achievement of PR or better to relapse or death due to MM (multiple myeloma)
DOR in Part B | from disease response to disease progression, assessed up to approximately 24 months
  DOR as assessed by local investigator:
  * The time from the first documented disease response after infusion of CR or better to the date of the first documented progression as assessed by IMGW or death due to MM, for subjects with a response of VGPR or PR to induction therapy, and
  * The time from the first documented disease response after infusion of PR or better to the date of the first documented progression as assessed by IMGW or death due to MM, for subjects with a response of VGPR or PR to induction therapy
Cmax of BCMA CAR-T cells | 24 months
  through qPCR-detected transgene of CART concentrations over time in peripheral blood and bone marrow
Tmax of BCMA CAR-T cells | 24 months
  through qPCR-detected transgene of CART concentrations over time in peripheral blood and bone marrow
AUC of BCMA CAR-T cells | 24 months
  through qPCR-detected transgene of CART concentrations over time in peripheral blood and bone marrow
Clast of BCMA CAR-T cells | 24 months
  through qPCR-detected transgene of CART concentrations over time in peripheral blood and bone marrow
number of patients with pre-existing and treatment induced immunogenicity (cellular and humoral) of BCMA CAR-T cell therapy | 24 Months

CONTACTS AND LOCATIONS:
Locations (8):
- United States (4):
  - Uni of Chi Medi Ctr Hema and Onco, Chicago, Illinois
  - Beth Israel Deaconess Medical Cente, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Novartis Investigative Site, Melbourne, Victoria, Australia
- Israel (2):
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Novartis Investigative Site, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No